CLINICAL TRIAL: NCT07286136
Title: Evaluation of The Cycle SyncingⓇ Method: A 12-Week Virtual Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLO LIVING, LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLOLIV202503
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Menstrual Cycle Disorder; Menstrual Symptoms; Hormonal Imbalance
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycle SyncingⓇ Intervention Group (Experimental): Participants will follow the Cycle SyncingⓇ Method daily for 12 weeks using the MyFLO app.
  Interventions: Dietary Supplement: MyFLO App

INTERVENTIONS:
Dietary Supplement: MyFLO App — Participants follow the Cycle SyncingⓇ Method using the MyFLO app daily for 12 weeks. This includes personalized food and workout plans, symptom logging, hormonal testing with MIRA devices (urine and BBT), continuous glucose monitoring (CGM), and weekly virtual coaching sessions.

SUMMARY:
This 12-week, 100% virtual single-group open-label trial evaluates the Cycle SyncingⓇ Method using the MyFLO app, MIRA hormonal monitoring, and continuous glucose monitoring to assess reduction in menstrual cycle symptom burden and hormonal regulation.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 22 - 42 years
* Regular menstrual cycles
* Willingness and ability to comply with daily app usage and device protocols
* Access to a compatible smartphone and reliable internet connection
* Ability to attend a weekly virtual call with study personnel

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Use of hormonal contraceptives or other medications known to alter menstrual cycle physiology
* Presence of significant comorbidities or chronic conditions that may interfere with study participation
* Any condition that, in the investigator's opinion, would make participation unsafe

Ages: 22 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Cycle Symptom Burden | Baseline, Month 1, Month 2, and Month 3
  Change in total symptom burden and severity scores as measured by validated symptom questionnaires.

SECONDARY OUTCOMES:
Time to Improvement in Symptom Burden | Baseline, Month 1, Month 2, and Month 3
  Time to statistically significant improvement in symptom burden, based on monthly assessments using validated questionnaires.
Change in Luteinizing Hormone (LH) levels | Baseline, Month 1, Month 2, Month 3
  Evaluation of changes in LH levels measured via the MIRA urine device.
Variations in Basal Body Temperature (BBT) | Baseline, Month 1, Month 2, Month 3
  Assessment of blood glucose trends throughout the study, with a focus on changes during the luteal phase of the menstrual cycle. Data will be collected continuously via CGM and analyzed monthly.
Impact on Blood Glucose Levels | Baseline, Month 1, Month 2, Month 3
  Assessment of blood glucose trends throughout the study, with a focus on changes during the luteal phase of the menstrual cycle.
Change in Estrone-3-glucuronide (E3G) levels | Baseline, Month 1, Month 2, Month 3
  Evaluation of changes in E3G levels measured via the MIRA urine device.
Change in Pregnanediol Glucuronide (PdG) levels | Baseline, Month 1, Month 2, Month 3
  Evaluation of changes in PdG levels measured via the MIRA urine device.
Change in Follicle-Stimulating Hormone (FSH) levels | Baseline, Month 1, Month 2, Month 3
  Evaluation of changes in FSH levels measured via the MIRA urine device.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States